CLINICAL TRIAL: NCT07202923
Title: Effect of Preoperative Tamsulosin and Silodosin on Successful Insertion Ureteral Access Sheath and Reduce Ureteral Injury in Non-Prestented Patients During Retrograde Intrarenal Surgery (RIRS). Assessment of Factors for Successful Ureteral Access Sheath Insertion. Randomized Clinical Trial.
Brief Title: Effect of Preoperative Alpha-blockers on Successful Insertion Ureteral Access Sheath and Reduce Ureteral Injury in Non-prestented Patients During RIRS. Assessment of Factors for Successful Ureteral Access Sheath Insertion.
Status: Completed | Type: Observational
Sponsor: St. Luke's Clinical Hospital, Russia (Other)
Responsible Party: Principal Investigator, Mikheev Yury, urologist, St. Luke's Clinical Hospital, St. Luke's Clinical Hospital, Russia
Other Study IDs: №19/2
Record Dates: First submitted 2025-08-16; First posted 2025-10-02 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Urolithiasis; Ureteral Injury; Ureteral Access Sheath; Retrograde Intrarenal Surgery
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group I (Tamsulosin): Non-prestented patients receiving 0.4 mg of Tamsulosin daily for 7 days before RIRS.
- Group II (Silodosin): Non-prestented patients receiving 8 mg of Silodosin daily for 7 days before RIRS.
- Group III: Prestented patients
- Group IV: Control group (non-prestented patients)

SUMMARY:
The aim of the study is to evaluate the effect of preoperative taking alpha-blockers (tamsulosin or silodosin) on the success rate of ureteral access sheath (UAS) insertion and the degree of ureteral injury during RIRS in non-prestented patients.

The results showed that patients who received alpha-blockers had a higher rate of successful UAS insertion and a lower degree of ureteral injury compared to non-prestented patients. In addition, patients with a BMI greater than 25 kg/m² and those older than 59 years demonstrated a higher success rate of UAS insertion and lower degree of ureteral injury.

DETAILED DESCRIPTION:
Study Title:

Effect of Preoperative Tamsulosin and Silodosin on Successful Insertion Ureteral Access Sheath and Reduce Ureteral Injury in Non-Prestented Patients During Retrograde Intrarenal Surgery (RIRS). Assessment of factors for successful ureteral access sheath insertion. Randomized clinical trial.

Study Design:

Prospective, randomized, open-label, controlled trial with four parallel arms. Conducted from July 2021 to June 2024.

Study Center:

Department of Urology, St. Luke's Clinical Hospital, St. Petersburg, Russia

Study Population:

140 patients, divided into four equal groups of 35 people each: Group I (Tamsulosin): Non-prestented patients receiving 0.4 mg of Tamsulosin daily for 7 days before RIRS.

Group II (Silodosin): Non-prestented patients receiving 8 mg of Silodosin daily for 7 days before RIRS.

Group III: Prestented patients. Group IV: Control group (non-prestented patients)

Interventions:

All patients received antibiotic prophylaxis with third-generation cephalosporins 30 minutes before surgery.

RIRS was performed using disposable flexible ureteroscopes. The UAS diameter was 11/13 Fr. Thulium fiber laser was used for lithotripsy. Stone fragmentation was performed in dusting and fragmentation modes, with a total power not exceeding 20 W and a fiber thickness of 200 µm.

Statistical Analysis:

Data were analyzed using Shapiro-Wilk, Mann-Whitney U, Kruskal-Wallis, and chi-square tests with Bonferroni correction (SPSS v26, JMP Pro 17). Statistical significance was set at p<0.05.

Key Findings:

Comparable baseline characteristics (p>0.05)

Significantly higher UAS success rates:

Tamsulosin: 31 (88.57%)

Silodosin: 32 (91.43%)

Prestented: 33 (94.29%)

Control: 62.86% (p=0.0008)

Preoperative taking Silodosin significantly reduced degree ureteral injury (p=0.0253).

Patients receiving alpha-blockers experienced less postoperative pain compared to the control group (p<0.0001) and less inflammatory changes in blood tests compared to prestented patients (WBC: p=0.0002; CRP: p<0.0001)

Patients with BMI ≥ 25 kg/m² and age ≥ 59 years had a higher success rate of UAS insertion (p<0,0001).

Patients with BMI ≥ 25 kg/m² and age ≥ 59 years have a lower degree of ureteral injury (p<0,0001).

Conclusions:

Preoperative taking of alpha-blockers (Tamsulosin or Silodosin) increases the success of UAS insertion.

Silodosin reduces the degree ureteral injury. Patients taking alpha-blockers less postoperative pain and inflammatory changes in blood tests.

A BMI ≥ 25 kg/m² and age ≥ 59 years increase the success of UAS insertion and reduce degree of ureteral injury

Clinical Implications:

This study provides evidence supporting the use of alpha-blockers, particularly silodosin, for passive ureteral dilation prior to RIRS in non-prestented patients, potentially reducing compications and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Kidney stone size: ≤2 cm
* Stone density >1000 Hounsfield units
* Sterile urine culture

Exclusion Criteria:

* Congenital anomalies of the urinary tract
* Urinary tract infections
* Upper urinary tract obstruction
* Prior reconstructive surgeries on the upper urinary tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an interventional RCT. Population characteristics are described in Eligibility Criteria and Arms sections
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
successful of ureteral access sheath insertion | Intraoperative
  Proportion of patients with successful UAS insertion
degree of ureteral injury | Perioperative
  Assessed using the PULS scale.Post-Ureteral Lesion Scale. Grade 0: No injury - intact ureter with no visible damage. Grade 1: Superficial mucosal injury - minor abrasions or erosions without disruption of the ureteral wall.
  Grade 2: Partial thickness injury - damage involving part of the ureteral wall, without full-thickness perforation; may have localized bleeding.
  Grade 3: Full-thickness ureteral injury - perforation of the ureteral wall with urine leakage, but the injury is limited in size.
  Grade 4: Extensive ureteral damage - large perforation with significant tissue destruction.
  Grade 5: Complete transection or avulsion - full disruption with loss of ureteral tissue, typically requiring complex reconstructive surgery.
postoperative pain | 6, 24, and 48 hours postoperatively
  Patient-reported pain intensity. The Visual Analog Scale for Pain (VASP) is a widely used, validated tool for the subjective measurement of pain intensity. It consists of a straight line, typically 10 centimeters (100 millimeters) in length, anchored by two verbal descriptors: "no pain" at the zero end and "worst imaginable pain" at the opposite end.
  Participants rate their current pain level by marking a point along the line that corresponds to their perception of pain intensity. The distance from the zero point to the mark (measured in millimeters or centimeters) quantifies the pain intensity on a continuous scale from 0 to 10 (or 0 to 100).
Inflammatory markers | Baseline and 24 hours postoperatively
  Change in in blood Leukocyte count, 10⁹/L C- reactive protein , mg/l
Factors influencing successful ureteral access sheath insertion | Until the completion of the study, on average 1 year
  Multivariate analysis of factors influencing successful UAS insetion. BMI of the patient - kg/m² Age of the patient

SECONDARY OUTCOMES:
Postoperative complications | through study completion, an average of 1 year
  Complications graded by Clavien-Dindo classification
Operative time | Intraoperative (measured from start to end of procedure)
  total operative time

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's Clinical Hospital, Saint Petersburg, Outside U.S./Canada, Russia

IPD SHARING:
Plan to Share IPD: Undecided
We are currently finalizing our data sharing policy. All required individual participant data underlying the reported results will be made available for regulatory purposes immediately upon request, and may be shared with researchers following publication after de-identification, contingent on submission of a methodologically sound proposal and compliance with institutional and national privacy regulations

REFERENCES:
- See also: Complete study data is available upon formal request by email . All legitimate data inquiries will be processed in accordance with applicable privacy regulations. — https://mail.google.com/mail/u/0/?tab=rm&ogbl#inbox